CLINICAL TRIAL: NCT03487874
Title: Efficacy of the 8th Cervical Nerve Root Block During Interscalene Brachial Plexus Block for Arthroscopic Shoulder Surgery: Prospective Randomized Controlled Study
Brief Title: Efficacy of the C8 Nerve Root Block During Interscalene Block for Anesthesia of the Posterior Aspect of the Shoulder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daegu Catholic University Medical Center (Other)
Responsible Party: Principal Investigator, JongHae Kim, Associate Professor, Daegu Catholic University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR-18-018
Record Dates: First submitted 2018-03-22; First posted 2018-04-04 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Brachial Plexus Block; Shoulder Pain
Keywords: 8th cervical nerve root block
MeSH Terms: conditions — Shoulder Pain | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interscalene block with C8 root block (Experimental): The 5th to 8th cervical nerve root block under ultrasound guidance using 25 to 30 ml of 0.75% ropivacaine
  Interventions: Procedure: Interscalene block with C8 root block; Drug: 0.75% ropivacaine
- Conventional interscalene block (Active Comparator): The 5th to 7th cervical nerve root block under ultrasound guidance using 25 to 30 ml of 0.75% ropivacaine
  Interventions: Procedure: Conventional interscalene block; Drug: 0.75% ropivacaine

INTERVENTIONS:
Procedure: Conventional interscalene block — Under ultrasound guidance, the 5th to 7th cervical nerve roots are blocked.
  Arms: Conventional interscalene block
Procedure: Interscalene block with C8 root block — Under ultrasound guidance, the 5th to 8th cervical nerve roots are blocked.
  Arms: Interscalene block with C8 root block
Drug: 0.75% ropivacaine — Placement of 25 to 30 ml of 0.75% ropivacaine around the cervical nerve roots
  Other Names: Naropin

SUMMARY:
This study evaluates the effects of selective 8th cervical nerve root block during interscalene brachial plexus block on the relief of pain intensity upon the introduction of a posterior portal during arthroscopic shoulder surgery. The 5th to 7th cervical nerve roots will be blocked in half of participants, while the 5th to 8th cervical nerve roots will be blocked in the other half.

DETAILED DESCRIPTION:
By blocking only the 5th to 7th cervical nerve blocks, conventional interscalene brachial plexus block spares the 8th cervical and 1st thoracic dermatomes which innervate the posterior aspect of the shoulder. To visualize the shoulder joint space during shoulder arthroscopic surgery, the introduction of a posterior portal is essential. However, conventional interscalene brachial plexus block cannot effectively relieve the pain caused by its insertion due to sparing of the 8th cervical and 1st thoracic dermatomes. The addition of the 8th cervical nerve root block to conventional interscalene brachial plexus block decreases pain intensity upon the introduction of a posterior portal.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status 1 and 2
* Arthroscopic shoulder surgery under interscalene brachial plexus block

Exclusion Criteria:

* Patient refusal
* Contralateral hemidiaphragmatic paralysis or paresis
* Contralateral vocal cord palsy
* Severe pulmonary restrictive disease
* Coagulopathy
* Allergy to local anesthetics or history of allergic shock
* Difficulty communicating with medical personnel
* Peripheral neuropathy or neurologic sequelae on the operative limb

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2019-08-09 (Actual)

PRIMARY OUTCOMES:
Pain intensity upon the introduction of a posterior portal | 50 minutes after interscalene block
  0, 1, and 2 represent no pain, mild pain, and severe pain, respectively.

SECONDARY OUTCOMES:
Sensory blockade | 30 minutes after interscalene block
  C5 to T1 dermatomal blockade graded from 0 to 2 (0 = no cold sensation, 1 = reduced cold sensation, and 2 = normal cold sensation) by applying ice to the shoulder
Motor blockade | 30 minutes after interscalene block
  Motor blockade of the radial, ulnar, median, musculocutaneous, and axillary nerves graded from 0 to 2 (0 = complete block, 1 = partial block, and 2 = no block)
Ipsilateral hemidiaphragmatic blockade | Before interscalene block and 30 minutes after interscalene block
  Extent of a reduction in the amplitude of excursion of the diaphragm on the vertical axis of the M-mode wave under M-mode ultrasound evaluation
Horner's syndrome | Before interscalene block and 30 minutes after interscalene block
  The extent of a reduction in the ipsilateral pupil size measured by a pupillometer Presence or absence of ptosis
Pulmonary function test | Before interscalene block and 30 minutes after interscalene block
  Forced expiratory volume at one second (FEV1) and FEV1/forced vital capacity before and 30 minutes after the end of local anesthetic injection
Complications related with interscalene block | 24 hours
  Presence or absence of vascular puncture, local anesthetic systemic toxicity, pneumothorax, and paresthesia
Numerical pain rating score at admission to postanesthetic care unit | 5 minutes
  Numerical pain rating score ranging from 0 to 10 (0 = no pain, 10 = worst pain imaginable) at admission to postanesthetic care unit
Numerical pain rating score at discharge from postanesthetic care unit | 30 minutes
  Numerical pain rating score ranging from 0 to 10 (0 = no pain, 10 = worst pain imaginable) at discharge from postanesthetic care unit
Numerical pain rating score between 6 and 12 hours after surgery | 6 and 12 hours
  Numerical pain rating score ranging from 0 to 10 (0 = no pain, 10 = worst pain imaginable) between 6 and 12 hours after surgery
Numerical pain rating score 24 hours after surgery | 24 hours
  Numerical pain rating score ranging from 0 to 10 (0 = no pain, 10 = worst pain imaginable) 24 hours after surgery
Worst numerical pain rating score | 24 hours
  Worst numerical pain rating score ranging from 0 to 10 (0 = no pain, 10 = worst pain imaginable) during 24 hours after surgery
Postoperative hour when pain starts to be felt | 24 hours
  Time at regression of anesthesia which starts to cause postoperative pain during 24 hours after surgery
Patient's satisfaction about surgical anesthesia and postoperative analgesia | 24 hours
  Likert scale consisting of "very dissatisfied", "dissatisfied", "unsure", "satisfied", and "very satisfied"
Dose of postoperative analgesic use | 24 hours
  Cumulative dose of analgesic required for postoperative analgesia during 24 hours after surgery
Frequency of postoperative analgesic use | 24 hours
  Frequency of analgesic use during 24 hours after surgery
Dose of intraoperative analgesic use | 2 hours
  Cumulative dose of analgesic to supplement incomplete surgical anesthesia
Frequency of intraoperative analgesic use | 2 hours
  Frequency of analgesic use to supplement incomplete surgical anesthesia
Conversion into general anesthesia | 1 hour
  Number of patients whose regional anesthesia is converted into general anesthesia due to incomplete surgical anesthesia provided by the regional anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Jong Hae Kim, MD, Principal Investigator — Daegu Catholic University Medical Center
Locations (1):
- Daegu Catholic University Medical Center, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim E, Choi CH, Kim JH. Effects of C8 nerve root block during interscalene brachial plexus block on anesthesia of the posterior shoulder in patients undergoing arthroscopic shoulder surgery: study protocol for a prospective randomized parallel-group controlled trial. Trials. 2019 Aug 28;20(1):533. doi: 10.1186/s13063-019-3624-9. PMID 31455407